CLINICAL TRIAL: NCT05424783
Title: Expanding an Active Surveillance Cohort to Improve Survivorship for Men With Favorable Risk Prostate Cancer
Brief Title: MRI And GPS Informing Choices for Prostate Cancer Treatment (MAGIC)
Acronym: MAGIC
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: STU00215555
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genomic Prostate Score assay and multi-parametric MRI of the prostate: Men with newly diagnosed NCCN very low to favorable intermediate risk prostate cancer will be enrolled at their post biopsy urologist visit. Once enrolled, participants will have their prostate tissue sent off for their Genomic Prostate Score assay and men will undergo a prostate MRI to evaluate for potentially missed clinically significant prostate cancer. In a subsequent urologist visit, participants will choose their treatment choice. Men who choose active surveillance for their primary treatment choice will be monitored per clinical routine by PSA, digital rectal exam, and active surveillance prostate biopsy in 12-18 months. After month 6, men will be followed through their electronic medical records system to track adherence to their 12-18 month active surveillance prostate biopsy.
  Interventions: Other: Genomic Prostate Score assay and Multi-parametric magnetic resonance imaging study of the prostate

INTERVENTIONS:
Other: Genomic Prostate Score assay and Multi-parametric magnetic resonance imaging study of the prostate — The Genomic Prostate Score is a 17 gene relative expression assay used to predict the presence of adverse pathologic findings at radical prostatectomy. This test is used to determine appropriateness for active surveillance. Prostate MRI is a prostate imaging test that has been shown to improve the detection of clinically significant prostate cancer using a PI-RADS scoring system. It relies on T2-weighted imaging, diffusion weighted imaging, dynamic contrast enhancement, and apparent diffusion coefficient to differentiate prostate cancer from normal prostate parenchyma and prostatitis.
  Other Names: GPS assay + mp-MRI

SUMMARY:
The overarching goal is to prospectively recruit men considering active surveillance for treatment in the MAGIC (MRI And GPS Informing Choices for prostate cancer treatment) Cohort to provide meaningful data on active surveillance in Blacks and in men served in safety net hospitals. Recent studies highlight significant promise for multi-parametric magnetic resonance imaging of the prostate (MRI) and Genomic Prostate Score assay (GPS) as tools to help risk stratify men on active surveillance to identify men likely to harbor undetected aggressive disease in their prostate. Given the risk data provided by these modalities and the low adherence with monitoring common in men served in public hospitals, both tools may improve safety via improved patient selection and patient adherence with monitoring. The downside is that excessive testing may lead to too many false positives and unnecessary treatment. Two hundred men with very low to intermediate risk prostate cancer were randomized into the 2-arm ENACT Clinical trial from 2016-2019 to study the impact of the GPS assay on treatment choice. Overall, 104 men received GPS assay and 96 controls did not receive the assay (a confirmatory test) right after being newly diagnosed with favorable risk prostate cancer.

For Aim 1, 222 men will be recruited into the MRI And GPS Informing Choices for prostate cancer treatment (MAGIC) study and they will be given the GPS assay and multi-parametric MRI of the prostate to provide personalized risk data for having aggressive tumors in their prostate. Between the ENACT and MAGIC study, there will be 3 groups of men who will have received both GPS & MRI, GPS alone, or neither test and can compare the impact of having 0,1 or 2 confirmatory tests on patient's adherence to active surveillance monitoring protocols over 18 months. The analyses will elucidate whether 1 or 2 tests are needed to improve adherence to monitoring. Monitoring is vital for detecting tumor progression early and avoiding cancer metastasis and death.

In Aim 2, the MAGIC study cohort will be leveraged to determine the accuracy of the Genomic Prostate Score assay and the prostate imaging- reporting and data system (PIRADS) score from the MRI in predicting which tumors will progress in 18 months. Progression is defined as increased Gleason grade group (GG) or change in prostate digital rectal examination findings. This serves two purposes. It will allow doctors and patients to categorize the patient as safe or risky for active surveillance. Secondly, it will allow doctors to identify which men on active surveillance need to be followed with annual prostate biopsies and which men can have their biopsies deferred for 3-5 years to reduce the number of prostate biopsies and their morbidities.

Lastly in Aim 3, the participants will rank the importance of these tests among a multitude of clinical, social, financial and interpersonal influences on their cancer treatment choice. By tallying the patient rankings, one can identify the most critical decision making factors that can be used to encourage increased selection of active surveillance.

DETAILED DESCRIPTION:
Active surveillance (AS) avoids or delays prostate cancer (PCa) treatment side effects for survivors. Blacks and men of lower socioeconomic status (SES) under-utilize this monitoring approach. Previous work has demonstrated that Genomic Prostate Score assay (GPS) is accurate in detecting adverse pathology at radical prostatectomy in Black and White men eligible for AS. One small study showed that Genomic Prostate Score (GPS) can predict tumor progression in 3 years. ENACT was closed to enrollment in 2019 and there were 200 men eligible for AS of lower SES enrolled into a randomized clinical trial assessing the impact of the GPS on patient treatment choice. AS was chosen by 77% of the participants for primary treatment and 72.1% of them were Black. The ENACT cohort now represents the second largest cohort of Black men on AS (n=112) with a median follow-up of 3 years. Moreover, recruitment took place at a Veterans Administration hospital, a County hospital and a state-funded University medical center serving men from with low rates of private insurance and a range of health literacy levels, thus complementing the data available from most AS cohorts. The long term goal is to reduce PCa over-treatment by improving the safety and acceptability of AS for men at higher risk for aggressive PCa. Multiparametric MRI of the prostate (mpMRI) has similarly been shown to predict tumor progression and Hence, the study will assess the accuracy of GPS for tumor progression, assess the impact of GPS on adherence to AS monitoring, and identify factors affecting AS selection in men of lower SES.

Aim 1. Assess the accuracy of the Genomic Prostate Score in a Black-enriched cohort to identify disease progression while on Active Surveillance over 3 years.

Methods: 66 of the 140 men on AS were randomized to receive the GPS. GPS tests will be performed on the 74 control participants' biopsies and coordinators will track all of the men for tumor progression (increase in Gleason score) on first AS prostate biopsy (PB) at 12-18 months. Tumor progression will be coded as Yes/No and receiver operating characteristics will be calculated for GPS while controlling for National Comprehensive Cancer Network (NCCN) risk group, age and race.

Aim 2. Compare the degree of adherence with NCCN active surveillance protocol at 18 months in men initially randomized to the GPS Intervention vs. Control group.

Methods: 140 of 200 men elected AS for initial treatment (101 Black/39 non-Black). As of January 2020, 3 men were lost to follow up. The proportion of men completing their surveillance prostate biopsy (PB) will be assessed at 18 months and there will be an assessment of the median number of prostate specific antigen (PSA) tests and digital rectal exams (DREs) completed per year between the 66 men randomized to the GPS on AS and the 74 controls.

Aim 3. Identify the main barriers and facilitators to initial active surveillance selection in a Black-enriched population.

Methods: Aim 3 leverage the clinical trial data and participants. All participants will be administered a survey to identify which factors encouraged or discouraged them from choosing AS, including patient and tumor factors, urologist treatment and decision making preference, and the GPS assay. There will be measures for medical mistrust, social support, employment status, insurance status, transportation and financial concerns, interactions with other PCa patients, and fear of job loss, side effects, surgery or of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have NCCN very low to favorable intermediate risk prostate cancer.
* Participants must be diagnosed within 3 months prior to study enrollment.
* Participants must be male, age 40-76 years old.
* Participants must be willing to consider active surveillance for treatment.

Exclusion Criteria:

* Participants with less than 10 years life expectancy.
* Participants unable to complete standardized surveys.
* Participants with no access to the rectum for a transrectal ultrasound.
* Participants with a contraindication to magnetic resonance imaging (MRI).

Ages: 40 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender men
Study Population: The target population for this study is participants with newly diagnosed favorable risk prostate cancer who are eligible for active surveillance for Prostate Cancer.
Sampling Method: Probability Sample
Enrollment: 222 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of men who had an active surveillance prostate biopsy by 18 months | 18 months after diagnostic prostate biopsy
  The men in the MAGIC study who chose active surveillance that complete their active surveillance prostate biopsy by 18 months after their diagnostic prostate biopsy will be compared to men who chose active surveillance in the ENACT Clinical Trial who received GPS alone (ENACT intervention arm) or neither GPS nor prostate MRI (ENACT control arm).

SECONDARY OUTCOMES:
The proportion of men with reclassification within 18 months | 18 months after diagnostic prostate biopsy
  The proportion of men with reclassification within 18 months of Visit 1 will be compared between the three groups: ENACT Control, ENACT GPS Intervention, MAGIC cohort.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Northwestern University and University of Illinois at Chicago are committed to making databases from clinical protocols available to interested investigators. This is subject to appropriate safeguards regarding protection of subjects' personal data. The first level of access will be to the investigators who have been involved in the conduct of the study. A second level is to the university for financial concerns around intellectual property and patents. Data can be provided in aggregate or at an individual level as an analytic database. The preferred format is a SPSS or SAS data set. These data sets will not contain subject identifying information. Once the proposed study is complete and the primary manuscript has been published, both character and analytic databases will be archived.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 18 months after study completion
Access Criteria: Affiliated with a research institution and proof of human subjects research training.

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT05424783/SAP_000.pdf
  • Informed Consent Form (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/83/NCT05424783/ICF_001.pdf